CLINICAL TRIAL: NCT01231438
Title: An Open, Randomized, Crossover Phase 2 Pilot Study of Treatment of Stage 3B Renal Failure With Active Vitamin D or a Phosphate Binder to Evaluate the Effect on the FGF23 and PTH Levels.
Brief Title: Treatment of Early Stage Renal Failure With Active Vitamin D or a Phosphate Binder.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Helse Stavanger HF (Other Government)
Collaborators: Rikshospitalet University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SUS2010GOLA01; 2010-020415-36 (EudraCT Number)
Record Dates: First submitted 2010-10-29; First posted 2010-11-01 (Estimated); Last update posted 2012-11-09 (Estimated); Status verified 2012-11

CONDITIONS: Kidney Failure
Keywords: Renal failure stage 3B
MeSH Terms: conditions — Renal Insufficiency | interventions — Sevelamer; alfacalcidol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Renvela (Experimental): Treatment for 2 weeks
  Interventions: Drug: Renvela
- Etalpha (Experimental): Vit D Treatment for 2 weeks
  Interventions: Drug: Etalpha

INTERVENTIONS:
Drug: Renvela — 800mg t.i.d. over 2 weeks
  Other Names: Sevelamercarbonate
  Arms: Renvela
Drug: Etalpha — 0.25ug o.d. for 2 weeks
  Other Names: Alfakalsidol
  Arms: Etalpha

SUMMARY:
Patients with reduced renal function normally develop hyperparathyroidism, which in turn is associated with increased cardiovascular risk and de-calcification. Hyperparathyroidism may be enhanced by an increased level of FGF23 which is often seen in the early stage of renal failure. This pilot study will investigate the FGF23-lowering effect of early initiation of treatment with a phosphate binder versus active vitamin D in an open crossover design.

ELIGIBILITY:
Inclusion Criteria:

* Renal failure stage 3B
* 25(OH)vitamin D level above 50 nmol/l
* Age over 18 years
* Written consent

Exclusion Criteria:

* Major surgery during the previous 6 months
* Myocardial infarct during the previous 6 months
* Unstable heart failure
* Ongoing treatment for any malignancy
* History of frequent infections
* Pregnancy
* Ongoing treatment with steroids, lithium or biphosphonates

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2010-10; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
FGF23 serum level | Change over 2 weeks of treatment

SECONDARY OUTCOMES:
Calcium serum level | Change over 2 weeks of therapy
Phosphate serum level | Change over 2 weeks of therapy
CTX-1 serum level | Change over 2 weeks of therapy
PINP serum level | Change over 2 weeks of therapy
PTH serum level | Change over 2 weeks of therapy

CONTACTS AND LOCATIONS:
Overall Officials: Lasse Göransson, MD PhD, Principal Investigator — Helse Stavanger HF
Locations (2):
- Norway (2):
  - Oslo Universitetssykehus Rikshospitalet, Oslo
  - Stavanger University Hospital, Stavanger

REFERENCES:
- [Result] Bleskestad IH, Bergrem H, Hartmann A, Godang K, Goransson LG. Fibroblast growth factor 23 and parathyroid hormone after treatment with active vitamin D and sevelamer carbonate in patients with chronic kidney disease stage 3b, a randomized crossover trial. BMC Nephrol. 2012 Jun 28;13:49. doi: 10.1186/1471-2369-13-49. PMID 22742720
- [Derived] Natale P, Green SC, Ruospo M, Craig JC, Vecchio M, Elder GJ, Strippoli GF. Phosphate binders for preventing and treating chronic kidney disease-mineral and bone disorder (CKD-MBD). Cochrane Database Syst Rev. 2025 Jun 27;6(6):CD006023. doi: 10.1002/14651858.CD006023.pub4. PMID 40576086